CLINICAL TRIAL: NCT02042183
Title: A Multicentre, Randomised, Placebo-controlled, Double-blinded Study of the Efficacy, Safety, and Pharmacokinetics of Lubiprostone in Paediatric Subjects Aged ≥ 6 Years to < 18 Years With Functional Constipation
Brief Title: Lubiprostone in Children With Functional Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Sucampo AG (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAG/0211PFC-1131; 2013-004384-31 (EudraCT Number); EMEA-000245-PIP01-08 (Other: EMEA Paediatric Investigational Plan)
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Constipation - Functional
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Intervention Model Description: Placebo controlled
Who Masked: Participant, Investigator
Masking Description: While the care provider and outcomes assessor were also blinded, this was classified as a double-blind trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lubiprostone (Experimental): Participants receive lubiprostone twice daily (BID) up to 12 weeks
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): Participants receive placebo BID up to 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — 12 or 24 mcg soft capsules of lubiprostone for oral administration, depending on baseline weight and response during week 1
  Other Names: Amitiza
  Arms: Lubiprostone
Drug: Placebo — 0 mcg soft capsules of placebo for oral administration
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
Study to determine if children (6-17 years old) with functional constipation will respond to being treated with lubiprostone for 12 weeks.

DETAILED DESCRIPTION:
Dose administration details:

* Participants with a body weight <50 kg at baseline received Lubiprostone 12 mcg BID for 12 weeks. If the dose was safe but did not show any efficacy at Week 1, dosage was increased to 24 mcg BID.
* Participants with a body weight >50 kg at baseline received Lubiprostone 24 mcg BID for 12 weeks. If the dose was unsafe at Week 1, dosage was decreased to 12 mcg BID.

ELIGIBILITY:
Inclusion Criteria:

* Medically-confirmed diagnosis of Functional Constipation per Rome III Diagnostic Criteria for Childhood Functional Constipation
* At least 6 years of age but less than 18 years of age at the time of randomisation
* Only stable dose of selective serotonin re-uptake inhibitors (SSRIs), serotonin-specific reuptake inhibitor (SNRIs), or monoamine oxidase inhibitors (MAO) inhibitors are allowed if subject is taking antidepressants

Exclusion Criteria:

* Any gastrointestinal (GI) condition, other than constipation and/or irritable bowel syndrome (IBS), affecting GI motility or defecation
* Untreated faecal impaction at the time of screening
* Medical/surgical condition that might interfere with the absorption, distribution, metabolism, or excretion of the study medication

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 606 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (116):
- United States (87):
  - University of Alabama Pediatric Gastroenterology, Birmingham, Alabama
  - University of South Alabama Women's and Children's Hospital, Mobile, Alabama
  - Arizona Children's Center at Maricopa Medical Center, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Applied Clinical Research of Arkansas, Little Rock, Arkansas
  - WCCT Global, Costa Mesa, California
  - Loma Linda University Health Care, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, San Francisco, San Francisco, California
  - MCB Clinical Research, Colorado Springs, Colorado
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Emmerson Clinical Research, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Palmetto Professional Research, Hialeah, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Savin Medical Group Research Center, Miami Lakes, Florida
  - Digestive & Liver Center of Florida, Orlando, Florida
  - Nemours Childrens Clinic, Pensacola, Florida
  - Children's Center for Digestive Healthcare/GI Care for Kids, Atlanta, Georgia
  - Center For Children's Digestive Health, Park Ridge, Illinois
  - Methodist Medical Center, Peoria, Illinois
  - PediaResearch, LLC - Newburgh, Newburgh, Indiana
  - UnityPoint Health Des Moines/ Blank Children's Clinic, Des Moines, Iowa
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Heartland Research Associates, Wichita, Kansas
  - University of Louisville Research Foundation Inc. Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - PediaResearch, LLC - Owensboro, Owensboro, Kentucky
  - Children's Hospital, New Orleans, Louisiana
  - Willis-Knighton Physician Network, Shreveport, Louisiana
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Virgo-Carter Pediatrics, Silver Spring, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Pioneer Clinical Research, Bellevue, Nebraska
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Digestive Diseases and Nutrition Center Women and Childrens Hospital of Buffalo, Buffalo, New York
  - Smart Medical Research, Inc., Jackson Heights, New York
  - NY Presbyterian Weill Cornell, New York, New York
  - Morgan Stanley Children's Hospital of New York Presbyterian, New York, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - PriMed Clinical Research, Beavercreek, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Square-1 Clinical Research, Inc., Erie, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children/Drexel University, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh UPMC, Pittsburgh, Pennsylvania
  - AAPRI Clinical Research, Warwick, Rhode Island
  - Coastal Pediatric Associates - James Island, Charleston, South Carolina
  - Coastal Clinical Research, Charleston, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Coastal Pediatrics Associates - Mount Pleasant, Mt. Pleasant, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - The Jackson Clinic, P.C., Jackson, Tennessee
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Monroe Carell Junior Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Tech University Health Sciences Center, Amarillo, Texas
  - Austin Center for Clinical Research, Austin, Texas
  - A1 Clinical Research, Baytown, Texas
  - 3rd Coast Research Associates, Corpus Christi, Texas
  - Childrens Medical Center Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Envision Clinical Research, LLC, Laredo, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Medical Clinics of Sealy, Sealy, Texas
  - Bridgerland Clinical Research, Logan, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Wee Care Pediatrics, Syracuse, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - INOVA Pediatric Digestive Diseases Center, Fairfax, Virginia
  - The Children's Hospital of the King's Daughter, Norfolk, Virginia
  - Pediatric Gastroenterology Carilion Medical Center, Roanoke, Virginia
  - Northwest Clinicial Research Center, Bellevue, Washington
  - Zain Research LLC, Richland, Washington
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - Universitair Kinderziekenhuis Brussel, Brussels
  - University Hospital Gasthuisberg, Leuven
  - CHC - Clinique Saint-Joseph, Montegnée
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - Centre de recherche du CHUS, Sherbrooke, Quebec
  - Sainte Justine University Health Center, Montreal
- France (4):
  - CHU-Bordeaux, Bordeaux
  - Groupe Hospitalier Est, Bron
  - Armand-Trousseau Teaching Hospital, Paris
  - Hôpital Necker, Paris
- Netherlands (4):
  - Emma Children's Hospital, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Maasstad Hospital Rotterdam, Rotterdam
  - Isala Klinieken, Zwolle
- Poland (8):
  - Medical University of Bialystok, Bialystok
  - Szpital Uniwersytecki, Bydgoszcz
  - ATOPIA Poradnie Specjalistyczne, Krakow
  - Medical University of Lodz, Lodz
  - Szpital Pediatryczny ICZMP, Lodz
  - Gabinet Lekarski Bartosc Korczowski, Rzeszów
  - Children's Memorial Health Institute, Warsaw
  - Przychodnia Specjalistyczna PROSEN, Warsaw
- United Kingdom (7):
  - Kent and Canterbury Hospital, Canterbury
  - Darlington Memorial Hospital, Darlington
  - Royal Hospital for Sick Children, Glasgow
  - Royal London Hospital, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Great Ormond Street Hospital for children NHS Foundation Trust, London
  - Sheffield Children Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No
Basic results are provided here, with statistical results and discussion reserved for publications.

REFERENCES:
- [Derived] Benninga MA, Hussain SZ, Sood MR, Nurko S, Hyman P, Clifford RA, O'Gorman M, Losch-Beridon T, Mareya S, Lichtlen P, Di Lorenzo C. Lubiprostone for Pediatric Functional Constipation: Randomized, Controlled, Double-Blind Study With Long-term Extension. Clin Gastroenterol Hepatol. 2022 Mar;20(3):602-610.e5. doi: 10.1016/j.cgh.2021.04.005. Epub 2021 Apr 7. PMID 33838349

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The two weeks between screening and treatment were used as a washout period for disallowed medications.
Groups:
- Lubiprostone: Participants receive lubiprostone twice daily (BID)
Period: Overall Study
Arm/Group | Lubiprostone | Placebo
Started | 404 | 202
Safety Population (All participants who took at least one dose of double-blinded study medication.) | 400 | 195
Modified Intent-to-treat (mITT) (All participants in safety population who have at least one efficacy assessment.) | 399 | 195
Completed | 339 | 166
Not Completed | 65 | 36
Not completed — Physician Decision | 7 | 2
Not completed — Lack of Efficacy | 4 | 3
Not completed — Non-compliance with Study Drug | 2 | 3
Not completed — Adverse Event | 17 | 6
Not completed — Other | 3 | 3
Not completed — Withdrawal by Subject | 21 | 16
Not completed — Site Terminated by Sponsor | 2 | 1
Not completed — Lost to Follow-up | 9 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Lubiprostone: Participants receive lubiprostone BID up to 12 weeks
- Total: Total of all reporting groups
Arm/Group | Lubiprostone | Placebo | Total
Number analyzed (Participants) | 404 | 202 | 606
Age, Customized [Count of Participants; unit: Participants] — Population: The modified intention-to-treat (mITT) population was used for reporting this baseline measure. The mITT population excluded participants from two sites that were terminated by the sponsor.
  Participants
    6-9 years: number analyzed (Participants) | 399 | 195 | 594
    6-9 years | 142 | 66 | 208
    10-13 years: number analyzed (Participants) | 399 | 195 | 594
    10-13 years | 153 | 78 | 231
    14-17 years: number analyzed (Participants) | 399 | 195 | 594
    14-17 years | 104 | 51 | 155
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The modified intention-to-treat (mITT) population was used for reporting this baseline measure. The mITT population excluded participants from two sites that were terminated by the sponsor.
  Participants
    number analyzed (Participants) | 399 | 195 | 594
    Female | 216 | 106 | 322
    Male | 183 | 89 | 272
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The modified intention-to-treat (mITT) population was used for reporting this baseline measure. The mITT population excluded participants from two sites that were terminated by the sponsor.
  Participants
    number analyzed (Participants) | 399 | 195 | 594
    Hispanic or Latino | 76 | 44 | 120
    Not Hispanic or Latino | 323 | 151 | 474
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The modified intention-to-treat (mITT) population was used for reporting this baseline measure. The mITT population excluded participants from two sites that were terminated by the sponsor.
  Participants
    number analyzed (Participants) | 399 | 195 | 594
    American Indian or Alaska Native | 0 | 3 | 3
    Asian | 3 | 3 | 6
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Black or African American | 67 | 39 | 106
    White | 308 | 138 | 446
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 20 | 11 | 31
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 7 | 12
  Netherlands | 14 | 32 | 46
  Belgium | 1 | 3 | 4
  United States | 174 | 348 | 522
  Poland | 3 | 8 | 11
  United Kingdom | 4 | 6 | 10
  France | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified as Overall Responders at Week 12
Description: An overall responder is defined as a participant who qualified as a weekly responder for 9 of the 12 treatment weeks, with durability demonstrated by at least 3 of the responder weeks occurring during the last 4 weeks of the treatment period. A weekly responder is defined as a participant who has at least 3 spontaneous bowel movements during the week, and at least one more than at baseline.
Time Frame: at Week 12
Population: mITT population
Measure: Count of Participants; unit: Participants
Groups:
- Lubiprostone: Participants receive lubiprostone BID for up to 12 weeks
- Placebo: Participants receive placebo BID for up to 12 weeks.
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 399 | 195
Participants | 76 | 28
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Other; p = 0.1609, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel (CMH) test stratified by baseline spontaneous bowel movement (SBM) frequency (<1.5 or ≥1.5)

2. Secondary Outcome: Mean Number of SBMs Observed Each Week for 12 Weeks
Description: Data provided is based on observed cases. Baseline is the average of the 2 weeks before being randomized. Participants are summarized by actual dose received after week 1.
Time Frame: within 12 Weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: Spontaneous bowel movements
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 399 | 195
Spontaneous bowel movements
  at Baseline | 1.40 (0.836) | 1.42 (0.855)
  at Week 1: number analyzed (Participants) | 387 | 186
  at Week 1 | 2.65 (2.137) | 2.50 (2.117)
  at Week 2: number analyzed (Participants) | 380 | 189
  at Week 2 | 2.68 (2.422) | 2.69 (2.328)
  at Week 3: number analyzed (Participants) | 371 | 184
  at Week 3 | 2.85 (2.446) | 2.59 (2.435)
  at Week 4: number analyzed (Participants) | 370 | 183
  at Week 4 | 2.94 (2.531) | 2.69 (2.499)
  at Week 5: number analyzed (Participants) | 356 | 175
  at Week 5 | 2.91 (2.498) | 2.68 (2.495)
  at Week 6: number analyzed (Participants) | 360 | 172
  at Week 6 | 2.91 (2.454) | 2.65 (2.163)
  at Week 7: number analyzed (Participants) | 342 | 172
  at Week 7 | 2.81 (2.483) | 2.75 (2.704)
  at Week 8: number analyzed (Participants) | 337 | 172
  at Week 8 | 2.94 (2.501) | 2.64 (2.444)
  at Week 9: number analyzed (Participants) | 336 | 165
  at Week 9 | 2.83 (2.286) | 2.37 (1.875)
  at Week 10: number analyzed (Participants) | 330 | 163
  at Week 10 | 2.68 (2.326) | 2.40 (2.103)
  at Week 11: number analyzed (Participants) | 328 | 163
  at Week 11 | 2.78 (2.251) | 2.60 (2.362)
  at Week 12: number analyzed (Participants) | 312 | 154
  at Week 12 | 2.90 (2.497) | 2.75 (2.530)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) in the safety population are reported for 14 weeks
Description: 1. Treatment-emergent adverse events are defined as any event with an onset date that is on or after the first dose of study medication and with an onset date no more than 7 days after the last dose of study medication.
  2. Participants are summarized in the dosing group assigned at randomization.
  The total number of participants in the 5% non-serious adverse event population was not provided, so the number affected is a total number of adverse events experienced by the 5% population.
Groups:
- Placebo: Participants received placebo BID for up to 12 weeks
Arm/Group | Lubiprostone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/400 | 0/195
Serious Adverse Events (participants affected / at risk) | 11/400 | 7/195
Other Adverse Events (participants affected / at risk) | 234/400 | 82/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lubiprostone (N=400) | Placebo (N=195)
Anaphylactoid reaction (Immune system disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 4 | 2
Suicidal ideation (Psychiatric disorders) | 1 | 1
Major depression (Psychiatric disorders) | 1 | 0
Hand-foot-and-mouth disease (Psychiatric disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Meniscus operation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lubiprostone (N=400) | Placebo (N=195)
Headache (Nervous system disorders) | 34 | 10
Nausea (Gastrointestinal disorders) | 57 | 14
Vomiting (Gastrointestinal disorders) | 45 | 12
Abdominal pain (Gastrointestinal disorders) | 42 | 23
Diarrhoea (Gastrointestinal disorders) | 28 | 6
Abdominal pain upper (Gastrointestinal disorders) | 20 | 6
Pharyngitis streptococcal (Infections and infestations) | 8 | 11

LIMITATIONS AND CAVEATS:
Outcome measures were not identified as such in the protocol, and some tables were recalculated at the request of the Food and Drug Administration, so revised data necessary to calculate the primary endpoint were posted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other